CLINICAL TRIAL: NCT00832130
Title: Randomized Clinical Trial for Treatment of Meibomian Gland Dysfunction and Evaporative Dry Eye
Brief Title: Treatment of Meibomian Gland Dysfunction and Evaporative Dry Eye
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TearScience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LF001
Record Dates: First submitted 2009-01-27; First posted 2009-01-29 (Estimated); Results first posted 2011-12-06 (Estimated); Last update posted 2011-12-12 (Estimated); Status verified 2011-12

CONDITIONS: Chalazion; Dry Eye Syndromes
MeSH Terms: conditions — Chalazion; Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Manual Mini System (Experimental): Treatment with experimental Manual Mini System
  Interventions: Device: Manual Mini System
- Warm Compress Therapy (Active Comparator): Control group receiving warm compress therapy in first study phase and crossover Manual Mini System treatment in second study phase
  Interventions: Device: Manual Mini System; Device: iHeat Portable Warm Compress Therapy

INTERVENTIONS:
Device: Manual Mini System — In-office device treatment for meibomian gland dysfunction by a physician
Device: iHeat Portable Warm Compress Therapy — At-home daily warm compress therapy
  Arms: Warm Compress Therapy

SUMMARY:
The objective of this study is to evaluate the clinical utility, safety and effectiveness of the Manual Mini System compared to standardized warm compress therapy for application of controlled, localized heat therapy in adult patients with chronic cystic conditions of the eyelids, including meibomian gland dysfunction, also known as evaporative dry eye or lipid deficiency dry eye, and chalazia.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age.
* Meibomian gland obstruction
* Dry eye symptoms
* Willingness to comply with study procedures and return for all visits

Exclusion Criteria:

* Ocular surgery, injury, or herpes infection within past 3 months
* Active ocular infection
* Active ocular inflammation or recurrent inflammation within past 3 months
* Moderate to severe allergic conjunctivitis
* Severe eyelid inflammation
* Eyelid abnormalities that affect lid function
* Ocular surface abnormalities that may compromise corneal integrity
* Macular disease
* Systemic disease condition or medication that causes dry eye
* Use of other treatments for meibomian gland dysfunction or dry eye
* Pregnant or nursing women
* Participation in another ophthalmic clinical trial within past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2009-02; Primary Completion 2009-06 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christy Stevens, OD, Study Director — TearScience, Inc.
Locations (11):
- United States (11):
  - Fayetteville, Arkansas
  - Morrow, Georgia
  - Highland Park, Illinois
  - Edgewood, Kentucky
  - Lexington, Kentucky
  - Winchester, Massachusetts
  - Jackson, Michigan
  - Bloomington, Minnesota
  - Stillwater, Minnesota
  - Charlotte, North Carolina
  - Lancaster, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 139 subjects (278 eyes) were enrolled at nine clinical sites between 03/04/2009 and 05/14/2009.
Pre-assignment Details: At the 2 Week visit, Control subjects stopped the warm compress therapy and received a single Manual Mini (LipiFlow) crossover treatment.
Period: Overall Study
Arm/Group | Manual Mini System | Warm Compress Therapy
Started | 69 | 70
Completed | 69 | 70
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Manual Mini System | Warm Compress Therapy | Total
Number analyzed (Participants) | 69 | 70 | 139
Age Continuous [Mean (Standard Deviation); unit: Years] | 52.4 (14.6) | 54.4 (16.4) | 53.4 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 53 | 97
  Male | 25 | 17 | 42

OUTCOME MEASURES:

1. Primary Outcome: Meibomian Gland Assessment (Total Meibomian Gland Secretion Score)
Description: Evaluation of secretion characteristics from the gland orifices along the lower eyelid. Assessment was based on the grading scale: 3 (clear liquid secretion), 2 (cloudy liquid secretion), 1 (inspissated), 0 (no secretion). The total meibomian gland secretion score was the sum of the grades for all 15 glands with a range of 0 to 45.
Time Frame: Baseline, 2 Weeks and 4 Weeks
Population: Results presented are for the Per Protocol population. 4 Weeks data for the Warm Compress Control group are after crossover.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Units Other Than Participants: Eyes
Arm/Group | Manual Mini System | Warm Compress Therapy
Number analyzed (Participants) | 65 | 68
Number analyzed (Eyes) | 130 | 136
Scores on a scale
  Baseline (N=130, 136) | 6.3 (3.5) | 5.6 (3.9)
  2 Weeks (N=130, 136) | 14.3 (8.7) | 6.1 (5.6)
  4 Weeks (N=128, 132) | 16.7 (8.7) | 11.7 (7.3)

2. Primary Outcome: Incidence of Device-related Adverse Events
Description: Number of eyes for which a device-related AE occurred
Time Frame: Baseline through 4 Weeks
Population: Results presented are of the Intent to Treat Population.
Measure: Number; unit: Events
Units Other Than Participants: Eyes
Arm/Group | Manual Mini System | Warm Compress Therapy
Number analyzed (Participants) | 69 | 70
Number analyzed (Eyes) | 138 | 140
Events | 4 | 2

3. Secondary Outcome: Dry Eye Symptoms (Total SPEED Score)
Description: Standard Patient Evaluation of Eye Dryness questionnaire. Assessment of subjects' frequency and severity of dry eye symptoms. The total score was calculated as the sum scores for all symptoms over a range of 0 to 28. A lower total SPEED score represents less frequent and/or less severe symptoms.
Time Frame: Baseline, 2 Weeks and 4 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Units Other Than Participants: Eyes
Arm/Group | Manual Mini System | Warm Compress Therapy
Number analyzed (Participants) | 65 | 68
Number analyzed (Eyes) | 130 | 136
Scores on a scale
  Baseline (N=130, 136) | 14.3 (4.8) | 14.8 (4.8)
  2 Weeks (N=130, 136) | 8.1 (5.5) | 11.2 (5.4)
  4 Weeks (N=128, 132) | 7.6 (5.8) | 7.9 (5.6)

4. Secondary Outcome: Ocular Surface Staining (Corneal Staining Sum Score)
Description: Corneal staining score in five corneal regions, evaluated on a scale from 0 (none), 1 (mild), 2 (moderate) to 3 (severe). The sum of the five corneal staining scores was on a scale from 0 to 15. A lower grade indicates less corneal surface desiccation.
Time Frame: Baseline through 4 Weeks
Population: Results presented are of the Intent to Treat Population. 4 Weeks data for the Control group are after treatment crossover.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Units Other Than Participants: Eyes
Arm/Group | Manual Mini System | Warm Compress Therapy
Number analyzed (Participants) | 69 | 70
Number analyzed (Eyes) | 138 | 140
Scores on a scale
  Baseline | 2.2 (2.2) | 2.0 (2.0)
  2 Weeks | 1.9 (2.0) | 2.0 (2.2)
  4 Weeks | 1.5 (1.7) | 1.6 (1.9)

5. Secondary Outcome: Intraocular Pressure
Description: Intraocular pressure (IOP) was evaluated by Goldmann applanation tonometry. Change in IOP from Baseline was assessed to confirm safety.
Time Frame: Baseline through 4 Weeks
Population: Results presented are of the Intent to Treat population. Post-Treatment results for the Control group are before crossover treatment. 4 Weeks results for the Control group are after crossover treatment.
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: Eyes
Arm/Group | Manual Mini System | Warm Compress Therapy
Number analyzed (Participants) | 69 | 70
Number analyzed (Eyes) | 138 | 140
mmHg
  Baseline (N=138, 140) | 13.3 (3.3) | 14.0 (2.8)
  Immediate Post-Treatment (N=138, 140) | 14.3 (3.3) | 15.0 (3.3)
  4 Weeks (138, 136) | 12.5 (2.9) | 13.1 (2.5)

6. Secondary Outcome: (LogMAR) Best Spectacle Corrected Visual Acuity
Description: Measurement of BSCVA at a distance using a logMAR chart under standard illumination. The logMAR ranged from -0.30 to 1.0. A lower logMAR value is a better visual acuity.
Time Frame: Baseline, 2 Weeks and 4 Weeks
Population: Results presented are of the Intent to Treat population. 2 Weeks data for the Control group are after control treatment, but before crossover treatment. 4 Weeks data for the Control group are after crossover treatment.
Measure: Mean (Standard Deviation); unit: LogMAR
Units Other Than Participants: Eyes
Arm/Group | Manual Mini System | Warm Compress Therapy
Number analyzed (Participants) | 69 | 70
Number analyzed (Eyes) | 138 | 140
LogMAR
  Baseline (N=138, 140) | 0.00 (0.12) | 0.01 (0.12)
  2 Weeks (N=136, 136) | -0.02 (0.13) | 0.02 (0.13)
  4 Weeks (N=138, 136) | -0.02 (0.12) | -0.01 (0.13)

7. Secondary Outcome: Discomfort Evaluation (Discomfort/Pain Score)
Description: Subject-reported numeric score reflecting low or high intensity. Scores ranged from 0 to 10, with 0 being no discomfort or pain and 10 being intolerable pain.
Time Frame: Treatment and 1 Day
Population: Results presented are of the Intent to Treat population. Only the Manual Mini group underwent a 1 day assessment.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Units Other Than Participants: Eyes
Arm/Group | Manual Mini System | Warm Compress Therapy
Number analyzed (Participants) | 69 | 70
Number analyzed (Eyes) | 138 | 140
Scores on a scale
  During Treatment (N=138, 140) | 1.4 (1.4) | 0.1 (0.7)
  Immediate Post-Treatment (N=138, 140) | 0.2 (0.6) | 0.0 (0.2)
  1 Day (N=138) | 0.2 (0.7) | NA (NA) — The Control group was not assessed for discomfort at 1 day post-treatment. This assessment refers only to discomfort after treatment with the Manual Mini System.

8. Primary Outcome: Tear Break-up Time
Description: Tear break-up time measured under a slit lamp biomicroscope following instillation of fluorescein dye in the eye. Time was measured in seconds with a maximum of 20. Higher tear break-up time indicates better tear film stability.
Time Frame: Baseline, 2 Weeks and 4 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Seconds
Units Other Than Participants: Eyes
Arm/Group | Manual Mini System | Warm Compress Therapy
Number analyzed (Participants) | 65 | 68
Number analyzed (Eyes) | 130 | 136
Seconds
  Baseline (N=130, 136) | 5.5 (2.9) | 5.4 (3.5)
  2 Weeks (N=130, 136) | 6.9 (5.0) | 5.3 (3.5)
  4 Weeks (N=128, 132) | 7.4 (5.5) | 6.3 (4.7)

ADVERSE EVENTS:
Time Frame: The presence of adverse events was evaluated at all study visits, including unscheduled visits.
Arm/Group | Manual Mini System | Warm Compress Therapy
Serious Adverse Events (participants affected / at risk) | 1/69 | 1/70
Other Adverse Events (participants affected / at risk) | 0/69 | 0/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Manual Mini System (N=69) | Warm Compress Therapy (N=70)
Elective Knee Surgery (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — The AE was systemic and unrelated to the device and study procedures.
Stroke (Vascular disorders) | 0 (0) | 1 (1) — The AE was systemic and unrelated to the device and study procedures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No